CLINICAL TRIAL: NCT01140139
Title: Active Immunotherapy Against HIV During Highly Active Anti-retroviral Therapy Followed by Repeated Treatment Interruptions
Brief Title: Dermal HIV-1 Immunization During Anti-retroviral Therapy Followed by Repeated Treatment Interruptions
Acronym: Vac09
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swedish Institute for Infectious Disease Control (Other)
Collaborators: European Union (Other); The Swedish Research Council (Other Government); Läkare mot AIDS Forskningsfond (Unknown)
Responsible Party: Professor Eric Sandström, Karolinska Institute and South Hospital, Stockholm
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DermHIVImm
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2006-02

CONDITIONS: HIV-1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HIV DNA + Hydroxyurea (Experimental): 0.4 mg of DNA plasmids encoding HIV env A, B, C and Rev B, gag A, B and RT mut formulated in PEI and glucose was applied topically with the DermaPrep procedure six times during cycles of 7 weeks of active HAART. Every immunization cycle was followed by four weeks of therapy interruption. The patients also received 500 mg of hydroxyurea daily.
  Interventions: Biological: HIV DNA Vaccine
- HIV DNA (Experimental): 0.4 mg of DNA plasmids encoding HIV env A, B, C and Rev B, gag A, B and RT mut formulated in PEI and glucose was applied topically with the DermaPrep procedure six times during cycles of 7 weeks of active HAART. Every immunization cycle was followed by four weeks of therapy interruption.
  Interventions: Biological: HIV DNA Vaccine
- Placebo (Placebo Comparator): PEI and glucose was applied topically with the DermaPrep procedure six times during cycles of 7 weeks of active HAART. Every immunization cycle was followed by four weeks of therapy interruption.
  Interventions: Biological: HIV DNA Vaccine

INTERVENTIONS:
Biological: HIV DNA Vaccine — 0.4 mg of DNA plasmids encoding HIV env A, B, C and Rev B, gag A, B and RT mut formulated in PEI and glucose was applied topically with the DermaPrep procedure six times during cycles of 7 weeks of active HAART. Every immunization cycle was followed by four weeks of therapy interruption.

SUMMARY:
In this study, the investigators evaluated a therapeutic HIV-1 DNA vaccine administered with a novel topical application method to 12 chronically HIV-infected cART treated patients. The HIV DNA plasmids used in this study encode for envelope gp160 of HIV-1 subtypes A, B and C, rev B, Gag A and B and reverse transcriptase (RT) B. The patients were randomly assigned to three groups; group 1 (n=4) were immunized six times with 0.4 mg of HIV DNA plasmids topically, group 2 (n=4) were immunized six times with 0.4 mg of HIV DNA plasmids topically and treated with 500 mg of hydroxyurea daily until visit 10, group 3 (n=4) four patients received placebo. The immunization was performed during three cycles of 7 weeks of cART followed by four weeks of therapy interruption. After the last cycle of cART the patients were maintained on a definitive treatment interruption until CD4+ T cell counts dropped below 350/ mm3 at two time points. Cellular and humoral immune responses, viral load and CD4+ T a cell count was analysed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 60 years
2. Female, who is documented infertile or in menopause since at least 1 year, or male, who are willing not father a child for the duration of the study.
3. HIV infection detected by two serological and/or HIV plasma RNA tests
4. On HAART for at least 6 months with less than 50 copies/ml of plasma HIV-1 RNA at two determinations over 3 months
5. Current CD4 count above 400
6. CD4 count nadir >200
7. Viral isolate pre ART available is preferable but not mandatory
8. Willing to consider stopping HAART repeatedly.
9. Willing to conform to a low alcohol intake (maximum of one glass per day)
10. Able to tolerate didanosine and hydroxyurea
11. Willing to change their HAART to exclude NNRTI and stavudine
12. Able to give informed consent
13. Availability for follow-up for planned duration of the study

Exclusion Criteria:

1. Patients with ongoing infection(s) other than HIV.
2. Prior or current pancreatitis or history of alcohol abuse.
3. Ongoing neuropathy and history of more than grade 1 neuropathy.
4. History of mutations to more than one class of anti-retroviral drugs or switched drugs more than once due to failure.
5. Sun or solarium exposure at the immunizing sites one month before or during the trial.
6. Cortisone treatment, systemic or local at the immunizing sites, one month before or during the trial.
7. Patients with signs of autoimmune diseases
8. Patients with creatinine > 2mg/dl, Hb < 12g/dl, leukocytes < 3,000ul, platelets <150,000/ul and LFT > 5x upper limit of normal
9. Patients on any immune modulating or investigational drug
10. Anamnestic allergy to kanamycin, plasmid gene products

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2006-09; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety and feasibility
  The safety and feasibility of dermal HIV-1 DNA vaccination will be evaluated by recording all medical events. They will be graded as to their seriousness, severity and relationship to the immunization. Plasma HIV-1 RNA levels and T-cell levels will be closely monitored. In addition to this the patient's individual experience and quality of life will be assessed.

SECONDARY OUTCOMES:
Treatment effects
  To evaluate whether dermal HIV-1 DNA vaccination can prolong periods without treatment in HIV-infected individuals. This will be evaluated by structured treatment interruption with close monitoring of HIV viral load and CD4+ T cell counts

CONTACTS AND LOCATIONS:
Locations (1):
- South Hospital, Stockholm, Sweden